CLINICAL TRIAL: NCT05926479
Title: Validation And Turkish Cross-Cultural Adaptation of Treatment Expectation Questionnaire (TEX-Q) Tool
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Other Study IDs: IstanbulBUFC
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Physiotherapy Patients
Keywords: patient; expectation; validity; reliability
MeSH Terms: interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- physiotherapy patient
  Interventions: Other: Translating the Questionnaire into Turkish and Related Processes; Other: Validity; Other: Reliability

INTERVENTIONS:
Other: Translating the Questionnaire into Turkish and Related Processes — The first step is the translation from the original language to the other language. The ideal target in the translation phase is to use people who are familiar with the structure of the original language and who are familiar with the language. Two forward translation and one reverse translation methods will be applied after obtaining the written permission of the authors. After the completion of this phase, the terminological differences arising from the translators in the translation process from the original language to Turkish will be collected and discussed on the questions. The cultural adaptation study will be terminated by determining the equivalence between the Turkish version of the index and the English original. The final version of the questionnaire and the necessary changes will be arranged specific to the investigator's society and the authors of the original questionnaire will be consulted and the questionnaire will be finalized.
Other: Validity — The scale will be applied by face-to-face technique and convergent (moderate-high correlation with optimism measure) and distant (low correlation with depression and anxiety measures) validity will be evaluated.
Other: Reliability — The reliability of the materials will be tested with Cronbach alpha.

SUMMARY:
The general treatment expectations of patients play a significant role in determining the outcomes of the different treatments they undergo. When it comes to physiotherapy programs, these expectations act as non-specific treatment components, capable of triggering subjective psychological changes and eliciting mechanisms that resemble placebo effects. When theory-based, multidimensional measurement tools that evaluate patients' expectations from various treatments are examined, the Treatment Expectation Questionnaire (TEX-Q) questionnaire stands out. The aim of this study is to ensure the validity and reliability of the Turkish version of this form, which can be answered by every patient receiving various treatments, as an objective alternative and to be included among other treatment expectancy measurement tools.

DETAILED DESCRIPTION:
This study includes the translation of the form after obtaining the relevant permissions, examining the internal consistency of the Turkish version, explanatory and confirmatory factor analysis, convergent validity and test-retest reliability processes.

The Turkish version of TEX-Q was applied to 200 patients who applied to the clinic for physiotherapy in the examination of internal consistency and exploratory factor analysis of the questionnaire. For convergent validity, 46 independent participants answered the Turkish version of the TEX-Q, the Positivity Scale, and the Hospital Anxiety and Depression Scale. The test-retest reliability within a 2-weeks interval was analysed in 63 of patients seeking physiotherapy program.

ELIGIBILITY:
Inclusion Criteria:

* ages between 18-65
* who would receive physiotherapy for at least 2 weeks for any indication

Exclusion Criteria:

* insufficient level of Turkish
* having any mental problems that would prevent participation in the study
* receiving another applied treatment other than the physiotherapy program

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who apply to physiotherapy clinic and will receive treatment for any indication
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Treatment Expectancy Questionnaire | Baseline
  It is a 21-item questionnaire, originally called the Treatment Expectation Questionnaire, developed by Alberts et al. in 2020, in which treatment expectations for different treatments can be measured in general and comparatively. The participant is asked to mark the number between 0 and 10 that he thinks corresponds to the appropriate value for him. Treatment benefit (items 1-3), positive effect (items 4-6), adverse effects (items 7-9), negative effect (items 10-11), treatment improvement (items 12-13), and behavioral control (items 14). -15) subheadings. Items 7-11 are reverse coded. There are 6 additional items of previous treatment experience. The total score of the questionnaire for the first 15 items is 150.

SECONDARY OUTCOMES:
Positivity Scale | Baseline
  Positivity Scale, directly evaluate the positivity levels of individuals. The original form of the instrument has a five-degree likert-type assessment. The Positivity Scale consists of eight items, one of which is reversed (item 6).
Hospital Anxiety and DepressionScale | Baseline
  The aim of the scale is to determine the severity and severity of the patient by determining the patient's susceptibility to anxiety and depression. The test has a total of 14 questions. Seven of these questions measure anxiety (odd numbers) and the remaining seven measure depression (even numbers). The cut-off points were 10 for anxiety and 7 for depression. Accordingly, those above this score are considered at risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Beyoglu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided